CLINICAL TRIAL: NCT03494088
Title: Mycobiome Evaluation in Children With Autism & GI Symptoms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jane J Alookaran, Pediatric gastroenterology fellow, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-17-1015
Record Dates: First submitted 2018-03-22; First posted 2018-04-11 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Autism; Gastrointenstinal Symptoms
Keywords: Autism; Abdominal Pain
MeSH Terms: conditions — Autistic Disorder; Abdominal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Blood
  * Saliva
  * Stool
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children with Autism with gastrointestinal (GI) symtpoms
- Children with Autism without gastrointestinal (GI) symtpoms
- Healthy Children

SUMMARY:
This study's primary aim is to explore the potential differences in the gut mycobiome of children with autism spectrum disorder compared to otherwise healthy children. The secondary objective of this study is to evaluate whether the presence of specific species of fungi (e.g. Candida tropicalis, C. albicans, or Saccharomyces cerevisiae), in stool: 1) correlates with increased gastrointestinal symptoms; 2) correlates with evidence of increased behavioral problems (as assessed by the Aberrant Behavior Checklist or Social Responsiveness Scale-2); or 3) plays the same role as a constituent of commensal gut microflora as in normal controls. The scale indicates severity of social deficits in the autism spectrum as mild, moderate or severe. Additionally, the study aims to compare the fecal and oral fungi in these children because many fecal mycobiota are felt to originate in the oropharynx.

ELIGIBILITY:
Inclusion Criteria:

* for autistic children with GI symptoms: confirmed diagnosis of autism spectrum disorder (ASD) and its severity (DSM-5: 299.00) by Autism Diagnostic Interview (ADI-R), Social Communication Questionnaire (SCQ), and Autism Diagnostic Observation SChedule-2 (ADOS-2); substantial gastrointestinal symptoms (as indicated by score of greater than 7 on the Gastrointestinal Symptoms Severity Index)
* for autistic children without GI symptoms: confirmed diagnosis of autism spectrum disorder (ASD) and its severity (DSM-5: 299.00) by Autism Diagnostic Interview (ADI-R), Social Communication Questionnaire (SCQ), and Autism Diagnostic Observation SChedule-2 (ADOS-2)
* for controls: healthy children

Exclusion Criteria:

* severe sensory impairment
* brain injury
* major psychiatric illness (e.g., psychotic disorders that might interfere with assessment). (however, children with common psychological problems such as depression and attention deficit hyperactivity disorder will not be excluded, given that doing so would result in a sample of children with ASD that would be unrepresentative of the pediatric ASD population as a whole.)- children who appear genetically syndromic (based on exam in the pediatric GI clinic)
* taking immunosuppressive medications
* abnormal screening labs
* GI diseases
* allergy to antibiotics
* fever or a pre-existing adverse event monitored in the study
* known history of hepatitis B/C or HIV
* known pregnancy
* use of probiotics in the last 60 d
* use of oral antibiotics/anti-fungal during the previous 2 weeks
* indwelling catheters/prosthetic devices

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy subjects will be recruited from The University of Texas Health Science Center at Houston general pediatrics clinic and adolescent clinic.
  Children with autism are referred to The University of Texas Health Science Center at Houston general pediatrics clinic and adolescent clinic.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Fecal Mycobiome Composition as assessed by sequencing of fecal fungal species | day 1

SECONDARY OUTCOMES:
Presence of fungal species Candida tropicalis | day 1
Presence of fungal species Candida albicans | day 1
Presence of fungal species Saccharomyces cerevisiae | day 1
Gastrointentinal (GI) symptoms as assessed by the GI Symptoms Severity Index | day 1
Behavioral problems as assessed by the Aberrant Behavior Checklist (ABC) | day 1
Behavioral problems as assessed by the Social Responsiveness Scale-2 (SRS-2) | day 1
Oral Mycobiome Composition as assessed by sequencing of oral fungal species | day 1
Gut inflammation as assessed by fecal calprotectin levels | day 1
Antifungal immunity as assessed by serum dectin 1 levels | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States